CLINICAL TRIAL: NCT06843642
Title: The Development of Diagnosis and Prognosis Predictive Model for Peripheral Nerve Disease Using Big Data From Magnetic Resonance Neurography: A Multicenter Cohort Study（MRN-PND）
Brief Title: The Development of Diagnosis and Prognosis Predictive Model for Peripheral Nerve Disease
Status: Completed | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Wuhan No.1 Hospital (Other); University Hospital Heidelberg (Other); West China Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0015-01
Record Dates: First submitted 2025-02-12; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Nerve Disease
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers
- Patients with Peripheral Nerve Disease

SUMMARY:
This is a retrospective observational cohort study (MRN-PND), aiming to explore the utility of contrast-enhanced MRN (ceMRN) compared to plain MRN in diagnosing peripheral nerve diseases and predicting the prognosis of patients with these conditions. Additionally, artificial intelligence (AI) methods are employed to enhance the diagnostic accuracy of MRN for peripheral nerve diseases and to precisely predict disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent MRN scanning at Wuhan Union Hospital between January 2015 and January 2025;
2. Age > 18 years;
3. Definitive clinical diagnosis (either healthy individuals or patients with a specific condition).

Exclusion criteria：

1. Poor quality of imaging;
2. Incomplete clinical data or loss to follow-up;
3. Unclear clinical diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy People and Patients with Peripheral Nerve Disease
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Correlation analysis of MR information and diagnosis outcome | 0.5 year
  The indicator is the area under the curve of the predict diagnosis outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital，Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei, China